CLINICAL TRIAL: NCT03795129
Title: Testing Utility of Commercially Available Sleep Trackers for Physician-Patient Communication Around Sleep Experience, Habits, and Behaviors
Brief Title: Testing Utility of Commercially Available Sleep Trackers for Physician-Patient Communication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regenstrief Institute, Inc. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Sleep Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Merck - 34
Record Dates: First submitted 2018-05-03; First posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Insomnia
Keywords: Early awakening
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized trial that is randomized at the clinic level.
Masking Description: Masking will not occur.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SleepLife Application w/FitBit (Experimental): Subject receives a FitBit. Subjects receive access to the SleepLife Application. Subjects receive training and assistance setting up use and access to the SleepLife Application.
  Subject physicians will receive subject sleep data. Subject and physicians have the option of messaging each other through the SleepLife application.
  Interventions: Behavioral: SleepLife Application w/FitBit
- FitBit w/Minimal to No SleepLife App. (Active Comparator): Subjects will receive a FitBit Subjects will be told about the SleepLife Application (but not be shown how to access it).
  Subjects will receive no training with regard to how to access SleepLife Application.
  Subjects' physicians will receive no subject sleep data.
  Interventions: Behavioral: FitBit w/Minimal to No SleepLife App.

INTERVENTIONS:
Behavioral: SleepLife Application w/FitBit — Subjects receive a FitBit. Subjects receive access to the SleepLife Application. Subjects receive training and assistance setting up use and access to the SleepLife Application.
  Subjects' physicians will receive subject sleep data. Subjects and physicians have the option of messaging each other through the SleepLife application.
  Arms: SleepLife Application w/FitBit
Behavioral: FitBit w/Minimal to No SleepLife App. — Subjects will receive a FitBit. Subjects will be told about the SleepLife Application (but not be shown how to access it).
  Subjects will receive no training with regard to how to access SleepLife Application.
  Subjects' physicians will receive no subject sleep data.
  Arms: FitBit w/Minimal to No SleepLife App.

SUMMARY:
Sleep related disorders are common in primary care practice. Sleep wear related data has not been utilized to improve sleep related communication between patients and providers. The study team is conducting a randomized study to improve physical-patient communication regarding sleep through a novel intervention based upon sleep wear and the Sleeplife® app.

DETAILED DESCRIPTION:
Based on a National US survey in 2012, 69% adults track at least one health indicator using either a tracking device or some other means. The main health indicators tracked were diet, weight, and exercise. Although not as extensive as the above health indicators, certain studies also looked at sleep indicators through the trackers to support validity of their use. Based on the study team's literature review, none of the studies looked at an intervention designed to utilize data-trackers-based data to improve physician-patient communication regarding sleep.

Commercially available and inexpensive exercise, fitness and sleep trackers are broadly available and consumer use is growing rapidly. Industry analysts estimate that over 30 million Americans have access to their sleep tracking data (e.g. Fitbit. Jawbone). Physicians seldom use patient-generated (i.e. subjective) sleep data (e.g. sleep diaries) and have been slow to integrate objective sleep data collected from commercial sleep trackers. Two commercial sleep trackers have been validated by independent testing. The National Sleep Foundation (NSF) has led recent efforts to establish normative data (i.e. appropriate ranges) for sleep duration and sleep quality. NSF, together with the Consumer Electronics Association (now Consumer Technology Association), has established a work-group involving over 40 sleep tracking technology companies which is working to standardize sleep tracking data collection and reporting. Finally, NSF has developed a tool ("SleepLife") that translates data retrieved from all commercially available sleep trackers into a personal sleep tracking record. This product has been tested rigorously for two years and publicly released in January 2016. These developments present the timely opportunity to test a new paradigm for patient and physician communication using objective patient data (sleep).

The study team will utilize a combination of observational and interventional study designs to achieve study objectives.

ELIGIBILITY:
Inclusion Criteria:

1. 18 and older
2. Have insomnia as identified by electronic record and/or a validated questionnaire
3. Prescription medication for insomnia with International Classification of Disease (ICD) codes: 327.*, 780.5*, 347.*; icd-10's G47* and medications: Ambien (zolpidem), Belsomra (suvorexant), Butisol (butabarbital), Doral (quazepam), Edluar (zolpidem), Estazolam, Flurazepam, Halcion (triazolam), Hetlioz (tasimelteon), Intermezzo (zolpidem), Lunesta (eszopiclone), Restoril (temazepam), Rozerem (ramelteon), Seconal (secobarbital), Silenor (doxepin), Sonata (zaleplon), and Zolpimist (zolpidem)

3. English speaking 4. Consentable in-person 5. Have access to a telephone with smart phone capabilities. (iOS/Android)

Exclusion Criteria:

1. Not English speaking
2. Have ischemic or hemorrhagic cerebrovascular disease affecting collection of study outcomes (via ICD codes I6*, 43*)
3. History of dementia (via ICD codes F0*, 290*)
4. History of Bipolar/Schizophrenia/Depression (via ICD codes F2*, F31*, 296*, 295*)
5. History of alcohol or substance abuse (via ICD codes F1*, 304*, 303*)
6. Incarcerated/Long Term Care (LTC)
7. Unable to complete study questionnaires due to hearing loss or blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-10 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of physicians using a commercially available sleep tracker assessed by the "Physician Satisfaction/Communication" questionnaire who saw an improvement in physician-patient dialogue regarding sleep and related behaviors and habits | Six Months
  For patient-physician communications from the physicians' end, the team will collect all scores, ranging from 1 to 5, for all the "Communication" questions in the "Physician Satisfaction/Communication" questionnaire. The scores will be summed up as the total communication score from physician, and the total score will be treated as continuous response variable. Then a binary variable indicating whether the physician is in the intervention (=1) or control (=0) arm will be treated as the main explanatory variable, a continuous variable regarding the time where the measurements are recorded, and the set of general demographic variables (age, race, gender, etc) will be used as covariates. We will use linear regression model, and select relevant variables using Bayesian information criterion (BIC) in a step-wise manner. The SleepLife app will be pulling time-to-sleep (TST), amount of time in minutes to sleep, number of awakenings greater than 5 minutes, and sleep efficiency.
Number of patient-physician communicationdialog assessed by using a commercially available sleep tracker assessed by the "Patient Satisfaction" questionnaire. | Six Months
  For patient-physician communications from the patients' end, the team will collect all the scores, ranging from 1 to 5, for all the "Communication" questions in the "Patient Satisfaction" questionnaire. The scores will be summed up as the total communication score from the patients' end, and the total score will be treated as continuous response variable. Then a binary variable indicating whether the patient is in the intervention (=1) or control (=0) arm will be treated as the main explanatory variable, a continuous variable regarding the time where the measurements are recorded, and the set of general demographic variables (age, race, gender, etc) will be used as covariates. Considering the linear responses and the cluster design, the team will use generalized estimating equation (GEE) model with an identity link function, and the team will select relevant variables using QIC in a step-wise manner.

SECONDARY OUTCOMES:
Number of physician subjects with satisfaction with sleep counseling that improves when presented with objective patient sleep data. | Six Months
  For physicians' satisfactory score, the team will collect all the scores, ranging from 1 to 5, for all the "GS" questions in the "Physician Satisfaction/Communication" questionnaire. The scores will be summed up as the total physicians' satisfaction score, and the total score will be treated as continuous response variable. Then a binary variable indicating whether the physician is in the intervention (=1) or control (=0) arm will be treated as the main explanatory variable, a continuous variable regarding the time where the measurements are recorded, and the set of general demographic variables (age, race, gender, etc) will be used as covariates. The team will use linear regression model, and select relevant variables using BIC in a step-wise manner.
Number of patients who feel that their communication with their physician has improved as a result of the program as measured by the "Patient Satisfaction" survey. | Six Months
  For patients' satisfaction, the team will collect all scores, ranging from 1 to 5, for all the "General Satisfaction" questions in the "Patient Satisfaction" questionnaire. These scores will be summed up as the total patients' satisfaction score for the treatment and interaction with the physician, as a result of the program. Then a binary variable indicating whether the patient is in the intervention (=1) or control (=0) arm will be treated as the main explanatory variable, a continuous variable regarding the time where the measurements are recorded, and the set of general demographic variables (age, race, gender, etc) will be used as covariates. Considering the linear responses and the cluster design, the team will use GEE model with an identity link function, and we will select relevant variables using QIC in a step-wise manner.

OTHER OUTCOMES:
To determine if data improves over time for measures related to total sleep time (TST) and satisfaction with sleep. | Six Months
  the team will collect all the scores, ranging from 0 to 100, for all the "Sleep Outcomes" questions in the sleep outcome questionnaire. These scores will be summed up as the total patients' sleep outcomes. Then a binary variable indicating whether the patient is in the intervention (=1) or control (=0) arm will be treated as the main explanatory variable, a continuous variable regarding the time where the measurements are recorded, and the set of general demographic variables (age, race, gender, etc) will be used as covariates. Considering the linear responses and the cluster design, we will use GEE model with an identity link function, and we will select relevant variables using QIC in a step-wise manner.

CONTACTS AND LOCATIONS:
Overall Officials: Babar Khan, MD, Principal Investigator — Regenstrief Institute, Inc.
Locations (1):
- Regenstrief Institute, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
The Regenstrief research team will use Protected Health Information (PHI) to conduct this study. Data that does not identify the subject will be shared with Merck Sharp & Dohme Corp. and the National Sleep Foundation. At this time, that is only the study visit day.

REFERENCES:
- [Result] Fox S, & Duggan M. Tracking for health. Pew Research Center, Pew Internet and American Life Project. 2013.
- [Result] Evenson KR, Goto MM, Furberg RD. Systematic review of the validity and reliability of consumer-wearable activity trackers. Int J Behav Nutr Phys Act. 2015 Dec 18;12:159. doi: 10.1186/s12966-015-0314-1. PMID 26684758
- [Result] de Zambotti M, Baker FC, Willoughby AR, Godino JG, Wing D, Patrick K, Colrain IM. Measures of sleep and cardiac functioning during sleep using a multi-sensory commercially-available wristband in adolescents. Physiol Behav. 2016 May 1;158:143-9. doi: 10.1016/j.physbeh.2016.03.006. Epub 2016 Mar 9. PMID 26969518
- [Result] de Zambotti M, Claudatos S, Inkelis S, Colrain IM, Baker FC. Evaluation of a consumer fitness-tracking device to assess sleep in adults. Chronobiol Int. 2015;32(7):1024-8. doi: 10.3109/07420528.2015.1054395. PMID 26158542
- [Result] Knutson KL, Phelan J, Paskow MJ, Roach A, Whiton K, Langer G, Hillygus DS, Mokrzycki M, Broughton WA, Chokroverty S, Lichstein KL, Weaver TE, Hirshkowitz M. The National Sleep Foundation's Sleep Health Index. Sleep Health. 2017 Aug;3(4):234-240. doi: 10.1016/j.sleh.2017.05.011. Epub 2017 Jun 20. PMID 28709508
- [Result] Hays, R.D., Davies, A.R., & Ware, J.E. (1987). Scoring the medical outcomes study patient satisfaction questionnaire: PSQ-III. MOS Memorandum.
- [Result] Campbell C, Lockyer J, Laidlaw T, Macleod H. Assessment of a matched-pair instrument to examine doctor-patient communication skills in practising doctors. Med Educ. 2007 Feb;41(2):123-9. doi: 10.1111/j.1365-2929.2006.02657.x. PMID 17269944
- [Result] Charlson ME, Sax FL, MacKenzie CR, Fields SD, Braham RL, Douglas RG Jr. Resuscitation: how do we decide? A prospective study of physicians' preferences and the clinical course of hospitalized patients. JAMA. 1986 Mar 14;255(10):1316-22. doi: 10.1001/jama.255.10.1316. PMID 3944949
- [Result] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Result] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Result] D'Hoore W, Sicotte C, Tilquin C. Risk adjustment in outcome assessment: the Charlson comorbidity index. Methods Inf Med. 1993 Nov;32(5):382-7. PMID 8295545
- [Result] Herr KA, Garand L. Assessment and measurement of pain in older adults. Clin Geriatr Med. 2001 Aug;17(3):457-78, vi. doi: 10.1016/s0749-0690(05)70080-x. PMID 11459715